CLINICAL TRIAL: NCT04212741
Title: Effectiveness of Oral Hyaluronic Acid (A+ HA(tm), TOP Pharm.) in Knee Osteoarthritis: Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Collaborators: TOP Pharm & Medicalware (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DMR101-IRB2-033
Record Dates: First submitted 2019-12-25; First posted 2019-12-30 (Actual); Last update posted 2020-01-03 (Actual); Status verified 2020-01

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A+ HA(tm) (Experimental): 20 ml oral solution of hyaluronic acid mixture in a bottle. Administration with 250~500 ml water under fasting condition in the morning.
  Interventions: Dietary Supplement: A+ HA(tm)
- Placebo (Placebo Comparator): 20 ml oral solution without active ingredients in a bottle. Administration with 250~500 ml water under fasting condition in the morning.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: A+ HA(tm) — oral solution of hyaluronic acid mixture
  Arms: A+ HA(tm)
Dietary Supplement: Placebo — oral solution with no-active ingredients
  Arms: Placebo

SUMMARY:
This is a double-blinded, placebo-controlled, randomized trial to assess the efficacy of oral solution of hyaluronic acid mixture (A+ HA(tm)). During 8 weeks treatment period, there were three follow-up visits requested (Week 2, Week 4 and Week 8).

DETAILED DESCRIPTION:
Subjects were initially screened at the Randomization/Baseline Visit (Week 0). Eligible subjects were randomized at the same visit into treatment period, and received the assigned treatment in a double-blind fashion for 8 weeks. Efficacy was measured by the several questionnaire including Knee injury and Osteoarthritis (KOOS), the Short Form-36 (SF-36) and Pittsburgh Sleep Quality Index (CPSQI) for each visit. Incidences of adverse events (AEs) were monitored for each subject once the subject had received 1 dose of study medication; the incidence of serious AEs (SAEs) were monitored for each subject once the subject had signed the informed consent through to the End-of-Study or ET Visit. Vital signs were measured at baseline and End-of-Study or ET Visit.

ELIGIBILITY:
Inclusion Criteria:

1. Age >= 40 years old
2. Male or Female
3. With osteoarthritis of the knee based on the definition of Ahlback 1968 and with significant symptoms within 30 days before enrollment.
4. No limitation for use of concomitant medication

Exclusion Criteria:

1. Use of Glucosamine within 1 month before enrollment
2. Osteoarthritis of the knee due to exercise or occupational injury
3. Allergy with Oral Hyaluronic Acid
4. Bilateral Total Knee Replacement
5. Pregnant
6. Need use wheelchairs
7. BMI≥40
8. With at least one condition: Known other causes of arthritis (infectious arthritis, rheumatoid arthritis, connective tissue disease, gout, pseudogout, or psoriatic arthritis), bony or soft tissue malignancy or skin lesions or peripheral neuropathy involving the lower extremities, cardiopulmonary disease which limits walking more than knee pain. Knee instability defined as report of knee bucking or locking within the past month of the study knee, major neurologic deficit that affects gait, psychiatric illness that limits informed consent, and parkinsonism.
9. Cancer

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score (KOOS) | 8 weeks
  A normalized score (0-100, 0 indicating extreme symptoms and 100 indicating no symptoms) was calculated.

SECONDARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | 8 weeks
  A normalized score (0-100, 0 indicating extreme symptoms and 100 indicating no symptoms) was calculated.
SF-36 | 8 weeks
  each item was recorded into score with a 0 to 100 range. Higher scores mean a better outcome.
Chinese version Pittsburgh Sleep Quality Index (CPSQI) | 8 weeks
  Total score of CPSQI from 0 (better) to 21 (worse) was used as the indicators of sleep quality

CONTACTS AND LOCATIONS:
Overall Officials: Shyu-Jye Wang, MD, Principal Investigator — China Medical University Hospital
Locations (1):
- TOP Pharm. & Medicalware, Taichung, Taiwan